CLINICAL TRIAL: NCT03779048
Title: Use of Pharmacotherapy to Improve Weight Loss in Early Non-responders to Behavioral Treatment
Brief Title: Use of Medication to Improve Weight Loss in Suboptimal Early Responders to Behavioral Treatment
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 832077
Record Dates: First submitted 2018-12-05; First posted 2018-12-19 (Actual); Results first posted 2025-03-11 (Actual); Last update posted 2025-03-11 (Actual); Status verified 2025-02

CONDITIONS: Obesity
Keywords: phentermine; Hypoglycemic agents; Incretins; Hormones; Appetitive Behavior; Appetite Depressants; Anti-Obesity Agents; Weight Loss; Body Weight; Body Weight Changes; Signs and Symptoms
MeSH Terms: conditions — Obesity; Appetitive Behavior; Anorexia; Weight Loss; Body Weight; Body Weight Changes; Signs and Symptoms | interventions — Behavior Therapy; Dosage Forms; Phentermine

STUDY DESIGN:
Intervention Model Description: Phase 1 is observational. Phase 2 is a double-blind, placebo-controlled, randomized controlled trial.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double-blind
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Phase 2: Behavioral Treatment + Placebo (Active Comparator): Participants with suboptimal early weight loss in the BT run-in will then be randomly assigned to 24 additional weeks of: 1) BT plus placebo (BT+P); or 2) BT plus medication (BT+M; phentermine 15.0 mg) in a double-blinded fashion. Both treatment groups will continue to attend individual BT sessions and will take a once daily study medication (placebo or phentermine 15.0 mg) for the duration of the intervention period.
  Early BT responders identified during the run-in will receive the same 24-week BT program, but will not receive study medication or be included in the randomized trial.
  Interventions: Behavioral: Behavioral Treatment; Drug: Placebo
- Phase 2: Behavioral Treatment + Medication (Active Comparator): Participants with suboptimal early weight loss in the BT run-in will then be randomly assigned to 24 additional weeks of: 1) BT plus placebo (BT+P); or 2) BT plus medication (BT+M; phentermine 15.0 mg) in a double-blinded fashion. Both treatment groups will continue to attend individual BT sessions and will take a once daily study medication (placebo or phentermine 15.0 mg) for the duration of the intervention period.
  Early BT responders identified during the run-in will receive the same 24-week BT program, but will not receive study medication or be included in the randomized trial.
  Interventions: Behavioral: Behavioral Treatment; Drug: Phentermine 15 MG
- Phase 1: 4-week Behavioral Treatment Run-in (Other): All enrolled participants will complete an initial 4-week behavioral treatment (BT) run-in. This run-in will be used to identify early non-responders to BT, defined by a weight loss <2% of initial weight after 4 weeks of BT. Early responders are those who lose >=2%.
  Only early non-responders will then be enrolled in the randomized trial.
  Interventions: Behavioral: Behavioral Treatment

INTERVENTIONS:
Behavioral: Behavioral Treatment — Behavioral treatment (BT) for weight loss includes diet and physical activity recommendations and behavior therapy strategies. All participants will complete an initial 4-week BT run-in, delivered in individual, 20-30 minute weekly sessions. After the end of the run-in, participants will be offered an additional 24 weeks of 20-30 minute individual BT sessions, occurring weekly for the first 12 weeks and every other week for the last 12 weeks (total of 18 visits).
  Other Names: Lifestyle modification; Behavioral weight loss
Drug: Placebo — The study medication (placebo or phentermine 15.0 mg) is a once-daily self-administered pill.
  Other Names: Placebo for medication
  Arms: Phase 2: Behavioral Treatment + Placebo
Drug: Phentermine 15 MG — The study medication (placebo or phentermine 15.0 mg) is a once-daily self-administered pill.
  Other Names: Medication
  Arms: Phase 2: Behavioral Treatment + Medication

SUMMARY:
This is a two-phase study. Phase 1 will evaluate obesity-related behavioral and biological characteristics as potential predictors of response to behavioral treatment (BT) for weight loss. Phase 2 is a double-blind, placebo-controlled, RCT to test whether adding weight loss medication to BT improves 24-week weight loss, as compared to BT with placebo, in subjects identified as having suboptimal early weight loss after 4 weeks of individual behavioral weight control. All participants, regardless of their early weight loss, will receive the same BT program of diet, physical activity, and behavior therapy for weight loss for an additional 24 weeks (28 total weeks of treatment).

DETAILED DESCRIPTION:
Subjects will be a total of 150 adults, aged 21-70 years, with a body mass index (BMI) of 31 kg/m2 or above (28 kg/m2 with an obesity-related comorbidity). In phase 1, eligible subjects will complete questionnaires and an in-person baseline assessment of obesity-related behavioral characteristics (satiety, hunger, the relative reinforcing value of food [RRVfood], and impulsivity [delay discounting]), neuropeptides, and gastric emptying. After this baseline assessment, participants will begin an initial 4-week behavioral treatment (BT) "run-in" delivered individually in 20-30 minute weekly sessions (delivered virtually).

The primary goal of phase 1 will be to evaluate baseline satiety, postprandial change in GLP-1, and gastric emptying as predictors of percent weight loss after 4 weeks of BT. We will also examine whether these variables predict categorization as a suboptimal early responder to BT (e.g., <2.0% loss; co-primary outcome).

Secondary endpoints of phase 1 are percent weight loss from the start of the BT run-in (week -4) to randomization (week 0) and categorization as a suboptimal early responder, as predicted by additional behavioral characteristics (hunger as measured by VAS ratings, RRVfood as measured using a computer task, and impulsivity as measured using a delay discounting computer task) and neuropeptides (higher fasting ghrelin, lower fasting leptin, and lower postprandial changes in insulin and PYY).

In phase 2, suboptimal early responders (based on weight loss during the BT run-in) will be randomly assigned to 24 weeks of: 1) BT plus placebo (BT+P); or 2) BT plus medication (BT+M; phentermine 15.0 mg). Both treatment groups will continue to attend 20-30 minute individual BT sessions (delivered virtually), weekly for the first 12 weeks and every other week for the last 12 weeks (total of 18 visits). Both treatment groups will also take once daily study medication (placebo or phentermine 15.0 mg) for the duration of the intervention period. Early BT responders identified during the run-in will receive the same 24-week BT program, but will not receive study medication or be included in the randomized trial.

The assessments administered at baseline - questionnaires, including behavioral testing, blood draws, and measurements of body weight - will be repeated at randomization (week 0) and at week 24.

The primary endpoint of phase 2 is change in body weight (i.e., % reduction in initial weight), as measured from randomization to week 24, among suboptimal early responders assigned to BT+P vs. BT+M. A randomized sample size of 50 non-responders (25 per group), assuming a 20% attrition rate, will give us 81.5% power to detect between-treatment group differences at week 24 of 4.5% (effect size: d = 0.82).

Secondary endpoints of phase 2 will include change in body weight in kg from randomization to week 24, as well as the portion of suboptimal early responders who achieve a post-randomization loss of ≥ 5% and ≥ 10% of initial body weight. We will also examine differences between suboptimal early responders treated with BT+M vs. BT+P in changes in hunger, satiety, the reinforcing efficacy of food, and impulsivity between randomization and week 24. A comparison will also be made in percent weight loss from randomization to week 24 between suboptimal early responders treated with BT+M and early responders treated with BT alone.

If you are interested in participating in this study, information and a link to contact the research team can be found here: https://clinicalresearch.itmat.upenn.edu/3XOX/ or you can call us at the numbers listed below.

ELIGIBILITY:
Inclusion Criteria:

1. BMI ≥ 31 kg/m² (or 28 kg/m2 with obesity-related comorbidity)
2. Age ≥ 21 years and ≤ 70 years
3. Eligible female patients will be:

   * non-pregnant, evidenced by a negative urine pregnancy test
   * non-lactating
   * surgically sterile or postmenopausal, or they will agree to continue to use an accepted method of birth control during the study. Acceptable methods of birth control are: hormonal contraceptives; double barrier method (condom with spermicide or diaphragm with spermicide); intrauterine device; surgical sterility; abstinence; and/or postmenopausal status (defined as at least 2 years without menses).
4. Subjects must:

   * have a primary care provider (PCP) who is responsible for providing routine care
   * understand and be willing to comply with all study-related procedures and agree to participate in the study by giving written informed consent
   * plan to remain in the Philadelphia area for the next 9 months or more

Exclusion Criteria:

1. Pregnant or nursing, or plans to become pregnant in the next 9 months.
2. Uncontrolled hypertension (systolic blood pressure ≥ 140 mm Hg or diastolic blood pressure ≥ 90 mm Hg)
3. Type 1 diabetes
4. Type 2 diabetes
5. A fasting blood glucose > 126 mg/dL (on second assessment after first elevated value)
6. History of cardiovascular disease (e.g., coronary artery disease, stroke, arrhythmias, congestive heart failure, or heart block greater than first degree
7. Clinically significant hepatic or renal disease
8. Hyperthyroidism
9. Other thyroid disease, not controlled
10. History of malignancy (except for non-melanoma skin cancer) in past 5 years
11. Narrow angle glaucoma
12. Presence or history of marked agitation
13. Current severe major depressive episode (BDI-II score ≥ 29), current active suicidal ideation, or history of suicide attempts within the past 5 years.
14. Any severity of thought or bipolar disorder, or bulimia nervosa.
15. Psychiatric hospitalization within the past 6 months
16. Self-reported alcohol or substance abuse within the past 6 months, including at-risk drinking (current consumption of ≥ 14 alcoholic drinks per week)
17. Past year history of drug abuse
18. Use in the past 2 weeks of monoamine oxidase inhibitors
19. Current use of serotonin-norepinephrine reuptake inhibitors (SNRIs; e.g. venlafaxine, duloxetine, desvenlafaxine, milnacipran, levomilnacipran).
20. Use in past 6 months of medications known to induce significant weight loss (i.e., prescription weight loss medications) or weight gain (e.g., chronic use of oral steroids, second generation antipsychotics)
21. Loss of ≥ 5% of initial body weight within the past 6 months
22. History of (or plans for) bariatric surgery (e.g., roux en y gastric bypass, sleeve gastrectomy, gastric banding), endoscopic intragastric balloon, or aspire assist.
23. Inability to walk 5 blocks comfortably or engage in some other form of aerobic activity (e.g., swimming)
24. Known or suspected allergy to sympathomimetic amines or related products
25. The receipt of any investigational drug within 6 months prior to this trial
26. Previous participation in this trial (e.g., randomized and failed to participate)
27. Changes to any chronic medication (type or dosage) within the past 3 months.
28. Any serious or unstable medical or psychological condition that, in the opinion of the investigator, would compromise the patient's safety or successful participation in the study

Other Therapy: Subjects will be expected to use medications (prescribed by their PCP) to control traditional cardiometabolic risk factors (e.g., hypertension, hypercholesterolemia, etc) and other co-morbid conditions, with the exception of medications listed above under "exclusions." In all cases, the subjects' PCP will be asked at the study's outset to keep medication does constant throughout the study, whenever possible. Subjects will be expected to have been on their medication regimen (including the dose) for 3 months prior to beginning the BT program.

To be eligible to participate in the randomized phase of the trial, subjects must also:

1. Complete at least 3 out of 4 treatment sessions during the 4-week BT run-in and attend a randomization visit. Attending an in-person makeup session within one week of a missed visit will count as having attended the run-in visit.
2. Lose < 2.0% of initial weight during the 4-week BT run-in.

Early BT responders who lose>=2% during the BT run-in will be offered the same 24-week BT program, but will not receive study medication or be included in the randomized trial.

Ages: 21 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 147 (Actual)
Dates: Start 2019-07-15 (Actual); Primary Completion 2022-05-25 (Actual); Study Completion 2022-05-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jena S Tronieri, PhD, Principal Investigator — Perelman School of Medicine at the University of Pennsylvania
Locations (1):
- University of Pennsylvania Center for Weight and Eating Disorders, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Tronieri JS, Ghanbari E, Chevinsky J, LaFata EM, Minnick AM, Rajpal S, Wang SY, Burcaw K, Berkowitz RI, Wadden TA. Anti-obesity medication for weight loss in early nonresponders to behavioral treatment: a randomized controlled trial. Nat Med. 2025 May;31(5):1653-1660. doi: 10.1038/s41591-025-03556-3. Epub 2025 Mar 7. PMID 40055520

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment occurred from July 2019 to November 2021. No participants could be enrolled between March 15, 2020 and July 1, 2020 due to COVID-19.
Pre-assignment Details: 147 pts consented & enrolled in phase 1. Of those, 16 did not enroll in phase 2: 7 did not complete >=3 BT sessions, 5 could not complete a randomization visit due to COVID-19, 3 were lost to follow-up and 1 declined.
  55 pts were early responders. For clinical purposes, these pts continued to receive BT for 24 weeks but because they were not eligible for randomization they were not part of the RCT.
  76 pts were early non-responders (4-week weight loss < 2%) randomized to BT+ placebo or BT+ med
Groups:
- Phase 1 (4-week Non-randomized BT run-in): The 147 participants that initially enrolled received 4 weeks of BT.
- Phase 2: Behavioral Treatment + Placebo: Participants with suboptimal early weight loss in the BT run-in will then be randomly assigned to 24 additional weeks of: 1) BT plus placebo (BT+P); or 2) BT plus medication (BT+M; phentermine 15.0 mg) in a double-blinded fashion. Both treatment groups will continue to attend individual BT sessions and will take a once daily study medication (placebo or phentermine 15.0 mg) for the duration of the intervention period.
  Early BT responders identified during the run-in will receive the same 24-week BT program, but will not receive study medication or be included in the randomized trial.
  Behavioral Treatment: Behavioral treatment (BT) for weight loss includes diet and physical activity recommendations and behavior therapy strategies. All participants will complete an initial 4-week BT run-in, delivered in individual, 20-30 minute weekly sessions. After the end of the run-in, participants will be offered an additional 24 weeks of 20-30 minute individual BT sessions, occurring weekly for the first 12 weeks and every other week for the last 12 weeks (total of 18 visits).
  Placebo: The study medication (placebo or phentermine 15.0 mg) is a once-daily self-administered pill.
- Phase 2: Behavioral Treatment + Medication: Participants with suboptimal early weight loss in the BT run-in will then be randomly assigned to 24 additional weeks of: 1) BT plus placebo (BT+P); or 2) BT plus medication (BT+M; phentermine 15.0 mg) in a double-blinded fashion. Both treatment groups will continue to attend individual BT sessions and will take a once daily study medication (placebo or phentermine 15.0 mg) for the duration of the intervention period.
  Early BT responders identified during the run-in will receive the same 24-week BT program, but will not receive study medication or be included in the randomized trial.
  Behavioral Treatment: Behavioral treatment (BT) for weight loss includes diet and physical activity recommendations and behavior therapy strategies. All participants will complete an initial 4-week BT run-in, delivered in individual, 20-30 minute weekly sessions. After the end of the run-in, participants will be offered an additional 24 weeks of 20-30 minute individual BT sessions, occurring weekly for the first 12 weeks and every other week for the last 12 weeks (total of 18 visits).
  Phentermine 15 MG: The study medication (placebo or phentermine 15.0 mg) is a once-daily self-administered pill.
Period: Phase 1: 4-week Non-randomized BT run-in
Arm/Group | Phase 1 (4-week Non-randomized BT run-in) | Phase 2: Behavioral Treatment + Placebo | Phase 2: Behavioral Treatment + Medication
Started | 147 | 0 (Phase not started yet) | 0 (Phase not started yet)
Completed | 134 (Three of these participants completed an assessment at the end of Phase 1 but were not eligible for Phase 2.) | 0 | 0
Not Completed | 13 | 0 | 0
Not completed — Lost to Follow-up | 8 | 0 | 0
Not completed — Could not complete visit due to COVID-19 | 5 | 0 | 0
Period: Phase 2: Randomized Trial
Arm/Group | Phase 1 (4-week Non-randomized BT run-in) | Phase 2: Behavioral Treatment + Placebo | Phase 2: Behavioral Treatment + Medication
Started | 0 (Phase completed) | 38 | 38
Completed | 0 | 36 | 36
Not Completed | 0 | 2 | 2
Not completed — Lost to Follow-up | 0 | 2 | 2

BASELINE CHARACTERISTICS:
Population: Baseline characteristics at the start of Phase 1 for all enrolled participants. Only 76 participants were identified as early non-responders and enrolled in the randomized trial.
Groups:
- Phase 1: 4-week Behavioral Treatment Run-in: All enrolled participants will complete an initial 4-week behavioral treatment (BT) run-in. This run-in will be used to identify early non-responders to BT, defined by a weight loss <2% of initial weight after 4 weeks of BT. Early responders are those who lose >=2%.
  Behavioral Treatment: Behavioral treatment (BT) for weight loss includes diet and physical activity recommendations and behavior therapy strategies. All participants will complete an initial 4-week BT run-in, delivered in individual, 20-30 minute weekly sessions. After the end of the run-in, participants will be offered an additional 24 weeks of 20-30 minute individual BT sessions, occurring weekly for the first 12 weeks and every other week for the last 12 weeks (total of 18 visits).
  Note: Data represent the baseline characteristics of all enrolled participants at the start of phase 1 (week -4). Only 76 participants were later eligible to enroll in the randomized trial.
Arm/Group | Phase 1: 4-week Behavioral Treatment Run-in
Number analyzed (Participants) | 147
Age, Continuous [Mean (Standard Deviation); unit: years] | 48.5 (12.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 128
  Male | 19
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 7
  Not Hispanic or Latino | 140
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 5
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 57
  White | 80
  More than one race | 4
  Unknown or Not Reported | 1
Weight (kg) [Mean (Standard Deviation); unit: kg] | 104.6 (19.8)
BMI (kg/m2) [Mean (Standard Deviation); unit: kg/m2] | 37.7 (6.4)

OUTCOME MEASURES:

1. Primary Outcome: Phase 1: Percent Weight Loss
Description: Co-primary outcomes - phase 1
Time Frame: Week -4 (start of BT run-in) to week 0 (randomization)
Population: Percent weight loss at the end of the 4-week BT run-in (phase 1) for all 134 individuals who provided a weight measurement at the end of the run-in (week 0) and for the subset of 76 individuals who were categorized as early non-responders and then enrolled in the randomized trial (phase 2)
Measure: Mean (Standard Deviation); unit: % change in weight
Groups:
- Phase 1: 4-week Behavioral Treatment Run-in: All enrolled participants will complete an initial 4-week behavioral treatment (BT) run-in. This run-in will be used to identify early non-responders to BT, defined by a weight loss <2% of initial weight after 4 weeks of BT. Early responders are those who lose >=2%.
  Only early non-responders will then be enrolled in the randomized trial.
  Behavioral treatment (BT) for weight loss includes diet and physical activity recommendations and behavior therapy strategies. All participants will complete an initial 4-week BT run-in, delivered in individual, 20-30 minute weekly sessions. After the end of the run-in, participants will be offered an additional 24 weeks of 20-30 minute individual BT sessions, occurring weekly for the first 12 weeks and every other week for the last 12 weeks (total of 18 visits).
- Behavioral Treatment + Placebo: All participants will complete an initial 4-week behavioral treatment (BT) run-in. Participants with suboptimal early weight loss in the BT run-in will then be randomly assigned to 24 additional weeks of: 1) BT plus placebo (BT+P); or 2) BT plus medication (BT+M; phentermine 15.0 mg) in a double-blinded fashion. Both treatment groups will continue to attend individual BT sessions and will take a once daily study medication (placebo or phentermine 15.0 mg) for the duration of the intervention period.
  Early BT responders identified during the run-in will receive the same 24-week BT program, but will not receive study medication or be included in the randomized trial.
  Behavioral Treatment: Behavioral treatment (BT) for weight loss includes diet and physical activity recommendations and behavior therapy strategies. All participants will complete an initial 4-week BT run-in, delivered in individual, 20-30 minute weekly sessions. After the end of the run-in, participants will be offered an additional 24 weeks of 20-30 minute individual BT sessions, occurring weekly for the first 12 weeks and every other week for the last 12 weeks (total of 18 visits).
  Placebo: The study medication (placebo or phentermine 15.0 mg) is a once-daily self-administered pill.
- Behavioral Treatment + Medication: All participants will complete an initial 4-week behavioral treatment (BT) run-in. Participants with suboptimal early weight loss in the BT run-in will then be randomly assigned to 24 additional weeks of: 1) BT plus placebo (BT+P); or 2) BT plus medication (BT+M; phentermine 15.0 mg) in a double-blinded fashion. Both treatment groups will continue to attend individual BT sessions and will take a once daily study medication (placebo or phentermine 15.0 mg) for the duration of the intervention period.
  Early BT responders identified during the run-in will receive the same 24-week BT program, but will not receive study medication or be included in the randomized trial.
  Behavioral Treatment: Behavioral treatment (BT) for weight loss includes diet and physical activity recommendations and behavior therapy strategies. All participants will complete an initial 4-week BT run-in, delivered in individual, 20-30 minute weekly sessions. After the end of the run-in, participants will be offered an additional 24 weeks of 20-30 minute individual BT sessions, occurring weekly for the first 12 weeks and every other week for the last 12 weeks (total of 18 visits).
  Phentermine 15 MG: The study medication (placebo or phentermine 15.0 mg) is a once-daily self-administered pill.
Arm/Group | Phase 1: 4-week Behavioral Treatment Run-in | Behavioral Treatment + Placebo | Behavioral Treatment + Medication
Number analyzed (Participants) | 134 | 38 | 38
% change in weight | 1.7 (1.6) | 0.9 (0.9) | 0.3 (1.1)

2. Primary Outcome: Phase 1: Number of Participants Who Are Categorized as Early Non-responders at Randomization (Week 0), Based on Percent Weight Loss
Description: Co-primary outcomes - phase 1
Time Frame: Week -4 (start of BT run-in) to week 0 (randomization)
Population: 16 were not enrolled in Phase 2: 7 did not complete at least 3 BT sessions 5 could not complete a randomization visit due to COVID-19 3 were lost to follow-up
  1 declined randomization
Measure: Count of Participants; unit: Participants
Groups:
- Original Enrolled Sample: 147 participants were enrolled in phase 1 (the 4-week behavioral treatment run-in)
Arm/Group | Original Enrolled Sample
Number analyzed (Participants) | 131
Participants | 76

3. Primary Outcome: Phase 1: Baseline Satiety, as Measured by Visual Analogue Scales (Range 0-100 mm) During a Test Meal; Satiety Quotient = [(Post-preload Rating - Fasting Rating Before Preload)] / (Energy Content of Preload in kcal) x 100.
Description: Primary predictor variable - phase 1
  Appetite suppression was first calculated as the average of 100 mm VAS items: hunger (reverse score), satisfaction, fullness, and prospective consumption (reverse score), such that higher scores indicate more appetite suppression (less appetite) for each test meal rating (fasting, then every 10m for 60m).
  The satiety quotient was then calculated for each post-preload rating using the above formula (see measure title). More positive scores show increased satiety (more appetite suppression). The final analysis uses the 60-minute area under the curve (AUC) for the satiety quotient to predict phase 1 weight loss outcomes. Area under the curve is calculated using the trapezoidal rule to sum the area under each 10-minute interval. AUC = Σ i = 0 to i = 60 10min*(x(i) + x(i-1))/2) where x is the satiety quotient value at time i. Higher scores indicate higher sustained satiety.
Time Frame: Baseline (week -5)
Population: mITT analysis was planned to include all participants who provided at least one post-baseline weight measurement (N=139 out of 147). Additional missing data were attributable to participants whose VAS responses at baseline were not complete enough to be scored.
Measure: Mean (Standard Deviation); unit: Satiety quotient*min
Arm/Group | Phase 1: 4-week Behavioral Treatment Run-in
Number analyzed (Participants) | 138
Satiety quotient*min | 787.3 (684.9)
Statistical Analysis 1: Comparison: Phase 1: 4-week Behavioral Treatment Run-in; Test type: Other — Regression using baseline scores to predict 4-week weight loss during the behavioral treatment run-in. Primary prediction analysis presented below was pre-specified to evaluate together postprandial satiety, postprandial increases in GLP-1 and gastric emptying (acetaminophen tests) and includes only the 125 participants from whom baseline blood samples could be obtained; p = .24, Regression, Linear; Controls for postprandial increases in GLP-1 and gastric emptying (acetaminophen tests); Standardized Beta coefficient = .11

4. Primary Outcome: Phase 1: Baseline Postprandial Change in GLP-1 During a Test Meal
Description: Primary predictor variable - phase 1.
  Blood samples were drawn at time 0 (fasting) and 30- and 60-min postprandial samples after consumption of a test meal. Value presented below is the 60-minute incremental area under the curve (AUC) for GLP-1 in picomoles (pM). Area under the curve is calculated using the trapezoidal rule to sum the area under each 0.5-hour interval. AUC = Σ i = 0 to i = 1 0.5hr*(x(i) + x(i-1))/2) where x is the GLP-1 value in pM at time i.
Time Frame: Baseline
Population: mITT analysis was planned to include all participants who provided at least one post-baseline weight measurement (N=139 out of 147). We could not include an additional 14 participants for whom we could not obtain at least one postprandial blood sample and/or a fasting blood sample.
Measure: Mean (Standard Deviation); unit: pM*hr
Arm/Group | Phase 1: 4-week Behavioral Treatment Run-in
Number analyzed (Participants) | 125
pM*hr | 0.52 (0.46)
Statistical Analysis 1: Comparison: Phase 1: 4-week Behavioral Treatment Run-in; Test type: Other — [test comment as in outcome 3, analysis 1]; p = .34, Regression, Linear; Controls for baseline postprandial satiety and gastric emptying (acetaminophen test); Standardized Beta coefficient = -0.09

5. Primary Outcome: Phase 1: Baseline Gastric Emptying During a Test Meal (Acetaminophen Test)
Description: Primary predictor variable - phase 1
  Gastric emptying was measured as the 60-minute area under the curve (AUC) for acetaminophen in micrograms per milliliter (ug/mL). Blood samples were obtained at time 0 (fasting/no acetaminophen - confirmatory) and 30 and 60-min after ingestion. Because acetaminophen is minimally absorbed by the stomach but quickly enters the bloodstream in the small intestine, gastric emptying is considered to be the primary factor influencing its appearance in the blood. Area under the curve is calculated using the trapezoidal rule to sum the area under each 0.5-hour interval. AUC = Σ i = 0 to i = 1 0.5hr*(x(i) + x(i-1))/2) where x is the acetaminophen value in ug/mL at time i.
Time Frame: Baseline
Population: mITT analysis was planned to include all participants who provided at least one post-baseline weight measurement (N=139 out of 147). We could not include an additional 13 participants for whom we could not obtain at least one postprandial blood sample.
Measure: Mean (Standard Deviation); unit: ug/mL*hr
Arm/Group | Phase 1: 4-week Behavioral Treatment Run-in
Number analyzed (Participants) | 126
ug/mL*hr | 5.22 (3.39)
Statistical Analysis 1: Comparison: Phase 1: 4-week Behavioral Treatment Run-in; Test type: Other — [test comment as in outcome 3, analysis 1]; p = .78, Regression, Linear; Controls for baseline postprandial satiety and postprandial change in GLP-1; Standardized Beta coefficient = 0.03

6. Primary Outcome: Phase 2: Percent Weight Loss
Description: Primary outcomes - phase 2 Percent change from randomization in body weight
Time Frame: Week 0 (randomization) to week 24
Measure: Mean (Standard Error); unit: % change in weight
Arm/Group | Behavioral Treatment + Placebo | Behavioral Treatment + Medication
Number analyzed (Participants) | 38 | 38
% change in weight | 2.8 (0.7) | 5.9 (0.7)
Statistical Analysis 1: Comparison: Behavioral Treatment + Placebo vs Behavioral Treatment + Medication; Test type: Superiority; p = .003, Mixed Models Analysis; Mean Difference (Final Values) = 3.1, 95% CI 2-sided [1.1 to 5.1], Standard Error of Mean 1.0

7. Secondary Outcome: Phase 1: Baseline Hunger, as Measured by Visual Analogue Scales (Range 0-100 mm, Higher = More Hunger) During a Test Meal
Description: Secondary predictor variable - phase 1
  Hunger was rated before and at 10 min intervals after a test meal for 60 min. Data presented below are the 60-min area under the curve (AUC) for postprandial change in hunger at baseline.(more negative = more sustained reduction in hunger). Area under the curve is calculated using the trapezoidal rule to sum the area under each 10-minute interval. AUC = Σ i = 0 to i = 60 10min*(x(i) + x(i-1))/2) where x is the hunger scale score at time i.
Time Frame: Baseline
Population: mITT analysis was planned to include all participants who provided at least one post-baseline weight measurement (N=139 out of 147).
Measure: Mean (Standard Deviation); unit: score on a scale*min
Arm/Group | Phase 1: 4-week Behavioral Treatment Run-in
Number analyzed (Participants) | 139
score on a scale*min | -770.97 (1272.98)
Statistical Analysis 1: Comparison: Phase 1: 4-week Behavioral Treatment Run-in; Test type: Other — Correlation between baseline postprandial hunger AUC and 4-week percent weight loss; p = .23, Regression, Linear; r = -.10

8. Secondary Outcome: Phase 1: Baseline Relative Reinforcing Value of Food (Computer Task), Number of Food Reinforcer Points Earned
Description: Secondary predictor variable - phase 1
  Subjects are allowed to work to earn points from a slot machine task at either of two computer stations, one of which provides points towards obtaining a serving of a preferred high-calorie food, and the other points towards a preferred low-calorie food. Points are earned on a progressive ratio scale that increases at fixed intervals. The primary outcome is the number of reinforcer points (servings) earned for the high energy density food, which is thought to reflect the subject's willingness to allocate time and effort to obtaining desired high-calorie foods. The minimum number of points that can be earned is 0; there is no specified maximum.
Time Frame: Baseline
Population: mITT analysis was planned to include all participants who provided at least one post-baseline weight measurement (N=139 out of 147). An additional 5 participants had missing data for this task at baseline.
Measure: Mean (Standard Deviation); unit: Points (portions) earned
Arm/Group | Phase 1: 4-week Behavioral Treatment Run-in
Number analyzed (Participants) | 134
Points (portions) earned | 1.85 (1.23)
Statistical Analysis 1: Comparison: Phase 1: 4-week Behavioral Treatment Run-in; Test type: Other — Correlation between baseline high energy density food reinforcer points earned and 4-week percent weight loss; p = .23, Regression, Linear; r = -.10

9. Secondary Outcome: Phase 1: Baseline Delay Discounting (Computer Task), Area Under the Curve Representing the Ratio of Immediate Reward Size to Time Delay
Description: Secondary predictor variable - phase 1
  Delay discounting is assessed via a computer program in which subjects are offered choices between small, immediate monetary rewards and larger, delayed rewards. The present delay discounting computer task used 7 time delays for $1000.
  The outcome is the area under the curve (AUC) representing the ratio of immediate reward size to time delay. AUCs were standardized to fall between 0 and 1 (Myerson et al., 2001) and were calculated for the plot of subjective values vs. delay, with lower values indicating greater discounting. Area under the curve is calculated using the trapezoidal rule to sum the area under each standardized time interval. AUC = Σ i = 0 to i = 1 proportion of max delay*(x(i) + x(i-1))/2) where x is the proportion of the maximum price inflection value at time i.
Time Frame: Baseline
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: dollar*day
Arm/Group | Phase 1: 4-week Behavioral Treatment Run-in
Number analyzed (Participants) | 139
dollar*day | 0.34 (0.23)
Statistical Analysis 1: Comparison: Phase 1: 4-week Behavioral Treatment Run-in; Test type: Other — Regression results using baseline AUC for delay discounting to predict 4-week percent weight loss, controlling for participant age; p = .033, Regression, Linear; r2 change = .033

10. Secondary Outcome: Phase 1: Baseline Implicit Wanting, Reaction Time on Leeds Food Preference Questionnaire
Description: Secondary predictor variable - phase 1
  Implicit wanting is measured by the Leeds Food Preference Questionnaire, a computer-based task using a forced choice paradigm for four categories: High-fat savory, high-fat sweet, low-fat savory, low-fat sweet. Reaction times are transformed to a standardized D-score that is then adjusted for the frequency of selection using a validated algorithm. Scores can range from -100 to 100 with more positive scores indicating a more rapid preference for one category over the other and more negative scores indicating the opposite.
Time Frame: Baseline
Population: mITT analysis was planned to include all participants who provided at least one post-baseline weight measurement (N=139 out of 147). We could not include an additional 2 participants due to their not completing the LFPQ at their baseline assessment
Measure: Mean (Standard Deviation); unit: Scale score
Arm/Group | Phase 1: 4-week Behavioral Treatment Run-in
Number analyzed (Participants) | 137
Scale score
  Implicit wanting of high-fat savory | 7.0 (26.9)
  Implicit wanting of high-fat sweet | -12.2 (27.7)
  Implicit wanting of low-fat savory | -13.5 (23.6)
  Implicit wanting of low-fat sweet | 18.7 (28.1)
Statistical Analysis 1: Comparison: Phase 1: 4-week Behavioral Treatment Run-in; Test type: Other — Correlation between baseline implicit wanting and 4-week percent weight loss. Because categories are scored relative to each other they cannot be included together in the same analysis, so separate correlations were conducted; p = .04, Regression, Linear — Correlation to Implicit wanting of High Fat Savory; r = .17
Statistical Analysis 2: Comparison: Phase 1: 4-week Behavioral Treatment Run-in; Correlation between baseline implicit wanting and 4-week percent weight loss. Because categories are scored relative to each other they cannot be included taughter in the same analysis, so separate correlations were conducted; Test type: Other — Correlation to Implicit wanting of Low Fat Savory; p = .72, Regression, Linear; r = -.03
Statistical Analysis 3: Comparison: Phase 1: 4-week Behavioral Treatment Run-in; Correlation between baseline implicit wanting and 4-week percent weight loss. Because categories are scored relative to each other they cannot be included together in the same analysis, so separate correlations were conducted; Test type: Other — Correlation to Implicit wanting of High Fat Sweet; p = .94, Regression, Linear; r = 0.01
Statistical Analysis 4: Comparison: Phase 1: 4-week Behavioral Treatment Run-in; [analysis description as in outcome 10, analysis 3]; Test type: Other — Correlation to Implicit wanting of Low Fat Sweet; p = .09, Regression, Linear; r = -0.15

11. Secondary Outcome: Phase 1: Baseline Fasting Ghrelin
Description: Secondary predictor variable - phase 1
  Blood samples were drawn at time 0 (fasting). Active ghrelin. Unit: Picograms per milliliter (pg/mL)
Time Frame: Baseline
Population: mITT analysis was planned to include all participants who provided at least one post-baseline weight measurement (N=139 out of 147). We could not include an additional 14 participants for whom we could not obtain a fasting blood sample or for whom fasting ghrelin results were out of range.
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Phase 1: 4-week Behavioral Treatment Run-in
Number analyzed (Participants) | 125
pg/mL | 75.65 (64.08)
Statistical Analysis 1: Comparison: Phase 1: 4-week Behavioral Treatment Run-in; Test type: Other — Correlation between baseline fasting active ghrelin and 4-week percent weight loss; p = .73, Regression, Linear; r = .03

12. Secondary Outcome: Phase 1: Baseline Fasting Leptin
Description: Secondary predictor variable - phase 1
  Unit: Picograms per milliliter (pg/mL) Blood samples were drawn at time 0 (fasting).
Time Frame: Baseline
Population: mITT analysis was planned to include all participants who provided at least one post-baseline weight measurement (N=139 out of 147). We could not include an additional 10 participants for whom we could not obtain a fasting blood sample or whose sample results were out of range.
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Phase 1: 4-week Behavioral Treatment Run-in
Number analyzed (Participants) | 129
pg/mL | 46980.6 (38772.3)
Statistical Analysis 1: Comparison: Phase 1: 4-week Behavioral Treatment Run-in; Correlation between baseline fasting leptin and 4-week percent weight loss; Test type: Other; p = .25, Regression, Linear; r = -.10

13. Secondary Outcome: Phase 1: Baseline Postprandial Change in Insulin During a Test Meal
Description: Secondary predictor variable - phase 1
  Blood samples were drawn at time 0 (fasting) and 30- and 60-min postprandial samples after consumption of a test meal. Incremental area under the curve in insulin measured in micro-international units per milliliter (ulU/mL). Area under the curve is calculated using the trapezoidal rule to sum the area under each 0.5-hour interval. AUC = Σ i = 0 to i = 1 0.5hr*(x(i) + x(i-1))/2) where x is the insulin value in ulU/mL at time i.
Time Frame: Baseline
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: ulU/mL*hr
Arm/Group | Phase 1: 4-week Behavioral Treatment Run-in
Number analyzed (Participants) | 125
ulU/mL*hr | 20.96 (13.08)
Statistical Analysis 1: Comparison: Phase 1: 4-week Behavioral Treatment Run-in; Test type: Other — Correlation between baseline postprandial AUC for change in insulin and 4-week percent weight loss; p = .72, Regression, Linear; r = -.03

14. Secondary Outcome: Phase 1: Baseline Postprandial Change in Peptide YY During a Test Meal
Description: Secondary predictor variable - phase 1
  Blood samples were drawn at time 0 (fasting) and 30- and 60-min postprandial samples after consumption of a test meal. Value presented below is the 60-minute incremental area under the curve (AUC) for PYY in picograms per milliliter (pgmL) at baseline. Area under the curve is calculated using the trapezoidal rule to sum the area under each 0.5-hour interval. AUC = Σ i = 0 to i = 1 0.5hr*(x(i) + x(i-1))/2) where x is the PYY value in pg/mL at time i.
Time Frame: Baseline
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: pg/mL*hr
Arm/Group | Phase 1: 4-week Behavioral Treatment Run-in
Number analyzed (Participants) | 125
pg/mL*hr | 7.44 (7.15)
Statistical Analysis 1: Comparison: Phase 1: 4-week Behavioral Treatment Run-in; Test type: Other — Correlation between baseline postprandial incremental AUC for PYY and 4-week percent weight loss; p = .82, Regression, Linear; r = -.02

15. Secondary Outcome: Phase 2: Weight Loss (kg)
Description: Secondary outcomes - phase 2
Time Frame: Week 0 (randomization) to week 24
Measure: Mean (Standard Error); unit: kg
Arm/Group | Behavioral Treatment + Placebo | Behavioral Treatment + Medication
Number analyzed (Participants) | 38 | 38
kg | 2.6 (0.7) | 5.7 (0.7)
Statistical Analysis 1: Comparison: Behavioral Treatment + Placebo vs Behavioral Treatment + Medication; Test type: Superiority; p = .002, Mixed Models Analysis; Mean Difference (Final Values) = 3.1, 95% CI 2-sided [1.1 to 5.0]

16. Secondary Outcome: Phase 2: Number of Participants With a Weight Loss of 5% or Greater of Randomization Body Weight at Week 24
Description: Secondary outcomes - phase 2
Time Frame: Week 0 (randomization) to week 24
Measure: Count of Participants; unit: Participants
Arm/Group | Behavioral Treatment + Placebo | Behavioral Treatment + Medication
Number analyzed (Participants) | 38 | 38
Participants | 8 | 20

17. Secondary Outcome: Phase 2: Number of Participants With a Weight Loss of 10% or Greater of Randomization Body Weight at Week 24
Description: Secondary outcomes - phase 2
Time Frame: Week 0 (randomization) to week 24
Measure: Count of Participants; unit: Participants
Arm/Group | Behavioral Treatment + Placebo | Behavioral Treatment + Medication
Number analyzed (Participants) | 38 | 38
Participants | 2 | 6

18. Secondary Outcome: Phase 2: Change in Appetite Suppression, as Measured by Visual Analogue Scales (Range 0-100 mm) During a Test Meal
Description: Secondary outcomes - phase 2
  Appetite suppression was first calculated as the average of 100 mm VAS items: hunger (reverse score), satisfaction, fullness, and prospective consumption (reverse score), such that higher scores indicate more appetite suppression (less appetite) for each test meal rating (fasting, then every 10m for 60m). The final analysis uses the 60-minute incremental area under the curve (AUC) for change in appetite suppression from fasting. Higher scores indicate higher sustained appetite suppression. Area under the curve is calculated using the trapezoidal rule to sum the area under each 10-minute interval. AUC = Σ i = 0 to i = 60 10min*(x(i) + x(i-1))/2) where x is the appetite suppression value at time i.
Time Frame: Week 0 (randomization) to week 24
Population: Randomized participants who completed the study (N = 71 of 76) and also completed the appetite test meal assessment at week 24 (N = 63 of 71). An additional two placebo-treated participants provided appetite ratings, but incremental area under the curve could not be calculated due to missing fasting item data.
Measure: Mean (Standard Deviation); unit: mm*min
Arm/Group | Behavioral Treatment + Placebo | Behavioral Treatment + Medication
Number analyzed (Participants) | 28 | 33
mm*min
  Randomization | 1167.7 (1124.8) | 1357.5 (1345.3)
  Week 24 | 862.8 (890.7) | 1245.3 (1072.9)

19. Secondary Outcome: Phase 2: Change in Hunger, as Measured by Visual Analogue Scales (Range 0-100 mm, Higher=More Hunger) During a Test Meal
Description: Secondary outcomes - phase 2
  Hunger was rated before and at 10 min intervals after a test meal for 60 min. Data presented below are the 60-min incremental area under the curve (AUC) for postprandial change in hunger at randomization and week 24. More negative scores indicate greater sustained reductions in hunger from fasting. Area under the curve is calculated using the trapezoidal rule to sum the area under each 10-minute interval. AUC = Σ i = 0 to i = 60 10min*(x(i) + x(i-1))/2) where x is the scale score at time i.
Time Frame: Week 0 (randomization) to week 24
Population: as for outcome 18
Measure: Mean (Standard Deviation); unit: mm*min
Arm/Group | Behavioral Treatment + Placebo | Behavioral Treatment + Medication
Number analyzed (Participants) | 28 | 33
mm*min
  Randomization | -1062.5 (1139.8) | -1113.2 (1294.6)
  Week 24 | -579.5 (1530.6) | -935.2 (1336.9)

20. Secondary Outcome: Phase 2: Change in Delay Discounting (Computer Task), Area Under the Curve Representing the Ratio of Immediate Reward Size to Time Delay
Description: Secondary outcomes - phase 2
  Delay discounting is assessed via a computer program in which subjects are offered choices between small, immediate monetary rewards and larger, delayed rewards. The present delay discounting computer task used 7 time delays for $1000.
  The outcome is the area under the curve (AUC) representing the ratio of immediate reward size to time delay. AUCs were standardized to fall between 0 and 1 (Myerson et al., 2001) and were calculated for the plot of subjective values vs. delay, with lower values indicating greater discounting. Area under the curve is calculated using the trapezoidal rule to sum the area under each standardized time interval. AUC = Σ i = 0 to i = 1 proportion of max delay*(x(i) + x(i-1))/2) where x is the proportion of the maximum price inflection value at time i.
Time Frame: Week 0 (randomization) to week 24
Population: Randomized participants who completed the study (N = 71 of 76) and also completed the delay discounting assessment at week 24 (N = 63 of 71).
Measure: Mean (Standard Deviation); unit: dollar*day
Arm/Group | Behavioral Treatment + Placebo | Behavioral Treatment + Medication
Number analyzed (Participants) | 30 | 33
dollar*day
  Randomization | 0.41 (0.30) | 0.38 (0.29)
  Week 24 | 0.42 (0.31) | 0.38 (0.25)
Statistical Analysis 1: Comparison: Behavioral Treatment + Placebo vs Behavioral Treatment + Medication; Test type: Superiority — Difference between placebo- and phentermine-treated participants in change in delay discounting area under the curve from randomization to week 24 was calculated using repeated measures ANCOVA, controlling for age; p = .68, ANCOVA; F = 0.17

21. Other Pre Specified Outcome: Phase 1: Baseline Eating Behavior as Measured by The Eating Inventory (EI); Dietary Restraint Subscale (Scored 0-21 Higher=More Restraint), Disinhibition Sub Scale (Scored 0-16 Higher=More Disinhibition), Hunger Sub Scale (Scored 0-14 Higher=More Hunger)
Description: Exploratory predictor variable - phase 1
  The Eating Inventory (EI); Dietary restraint subscale (scored 0-21 higher=more restraint), Disinhibition sub scale (scored 0-16 higher=more disinhibition), Hunger sub scale (scored 0-14 higher=more hunger)
Time Frame: Baseline
Population: mITT analysis was planned to include all participants who provided at least one post-baseline weight measurement (N=139 out of 147). Eating Inventory scores for an additional 4 participants could not be calculated due to missing items
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Phase 1: 4-week Behavioral Treatment Run-in
Number analyzed (Participants) | 135
score on a scale
  EI Dietary Restraint | 9.2 (3.7)
  EI Disinhibition | 8.9 (3.3)
  EI Hunger | 5.9 (3.3)
Statistical Analysis 1: Comparison: Phase 1: 4-week Behavioral Treatment Run-in; Test type: Other — Regression using the three Eating Inventory subscales (Cognitive restraint, disinhibition, hunger) to predict 4-week weight loss; p = .75, Regression, Linear — For full model including all 3 predictors; r2 = .01

22. Other Pre Specified Outcome: Phase 1: Baseline Appetite Ratings (Ratings of Appetite During the Past Week Using Visual Analogue Scales, Scored 0-100 mm, Higher=Greater Amount or Frequency)
Description: Exploratory predictor variable - phase 1
  Appetite was rated weekly using the Control of Eating Questionnaire. Participants were asked to rate items based on their appetite in the past week. For the present analysis, "appetite" was calculated as the mean of the ratings for hunger, fullness after meals (reversed), and thoughts about wanting food. Higher scores (Range 0 - 100) indicate greater past-week appetite.
Time Frame: Baseline
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Phase 1: 4-week Behavioral Treatment Run-in
Number analyzed (Participants) | 139
mm | 50.7 (12.0)
Statistical Analysis 1: Comparison: Phase 1: 4-week Behavioral Treatment Run-in; Test type: Other — Correlation between baseline past-week appetite and 4-week percent weight loss; p = .31, Regression, Linear; r = -.09

23. Other Pre Specified Outcome: Phase 1: Baseline Reinforcing Value of Food as Measured by the Power of Food Scale
Description: Exploratory predictor variable - phase 1 Power of Food Scale (PFS; range 1-5, higher=greater power of food)
Time Frame: Baseline
Population: mITT analysis was planned to include all participants who provided at least one post-baseline weight measurement (N=139 out of 147). We could not include an additional 6 participants due to missing items on the scale
Measure: Mean (Standard Deviation); unit: Scale score
Arm/Group | Phase 1: 4-week Behavioral Treatment Run-in
Number analyzed (Participants) | 133
Scale score | 2.7 (0.9)

24. Other Pre Specified Outcome: Phase 1: Baseline Sensitivity to Reward as Measured by the Behavioral Inhibition/Activation Scale (BIS/BAS)
Description: Exploratory predictor variable - phase 1
  BIS subscale range 7-28, higher = greater inhibition; BAS reward responsiveness sub scale range 5-20, higher=greater reward responsiveness
Time Frame: Baseline
Population: mITT analysis was planned to include all participants who provided at least one post-baseline weight measurement (N=139 out of 147). We could not include an additional 5 participants due to missing items on the BIS-BAS scale
Measure: Mean (Standard Deviation); unit: Scale score
Arm/Group | Phase 1: 4-week Behavioral Treatment Run-in
Number analyzed (Participants) | 134
Scale score
  BIS Total | 14.2 (4.0)
  BAS Reward | 8.2 (2.2)
Statistical Analysis 1: Comparison: Phase 1: 4-week Behavioral Treatment Run-in; Test type: Other — Regression using baseline scores for Behavioral Inhibition (BIS) and Behavioral Activation fro Reward to predict 4-week weight loss during the behavioral treatment run-in; p = .03, Regression, Linear; r2 = 0.05

25. Other Pre Specified Outcome: Phase 1: Baseline Impulsivity as Measured by The Barratt Impulsiveness Scale
Description: Exploratory predictor variable - phase 1
  BIS-15, range 15-60, higher= more impulsiveness
Time Frame: Baseline
Population: mITT analysis was planned to include all participants who provided at least one post-baseline weight measurement (N=139 out of 147). We could not include an additional 3 participants due to missing items on the BIS-15 scale
Measure: Mean (Standard Deviation); unit: Scale score
Arm/Group | Phase 1: 4-week Behavioral Treatment Run-in
Number analyzed (Participants) | 136
Scale score | 28.7 (6.5)
Statistical Analysis 1: Comparison: Phase 1: 4-week Behavioral Treatment Run-in; Test type: Other — Correlation between baseline BIS-15 total score and 4-week percent weight loss; p = .76, Regression, Linear; r = 0.03

26. Other Pre Specified Outcome: Phase 1: Baseline Binge Eating as Measured by The Questionnaire on Eating and Weight Patterns (QEWP-5); Measure Categorizes Participants Based on Whether They May Meet Diagnostic Criteria for Binge Eating Disorder
Description: The potential presence or absence of binge eating disorder (BED) is determined based on the participant's responses to questions assessing DSM-5 criteria for the disorder. Participants are categorized as potentially having BED, potentially having subthreshold BED (meets all criteria except frequency) or unlikely to have BED based on questionnaire responses.
  Exploratory predictor variable - phase 1.
Time Frame: Baseline
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 1: 4-week Behavioral Treatment Run-in
Number analyzed (Participants) | 131
Participants
  Potential BED | 17
  Potential subthreshold BED | 6
  Unlikely to have BED | 108

27. Other Pre Specified Outcome: Phase 1: Baseline Craving Frequency as Measured by the Food Craving Q Trait - Reduced
Description: Exploratory predictor variable - phase 1
  The Food Craving Q Trait - Reduced, total score (sum of 15 items, range 15-90); higher scores indicate more food cravings
Time Frame: Baseline
Population: mITT analysis was planned to include all participants who provided at least one post-baseline weight measurement (N=139 out of 147). We could not include an additional 3 participants due to missing items on the scale
Measure: Mean (Standard Deviation); unit: Scale score
Arm/Group | Phase 1: 4-week Behavioral Treatment Run-in
Number analyzed (Participants) | 136
Scale score | 42.9 (15.9)

28. Other Pre Specified Outcome: Phase 1: Baseline Emotional Eating as Measured by the Dutch Eating Behaviour Questionnaire (DEBQ)
Description: Exploratory predictor variable - phase 1
  The Dutch Eating Behaviour Questionnaire (DEBQ) Emotional Eating subscale, mean of 13 items, range 1-5, higher scores indicate more emotional eating
Time Frame: Baseline
Population: as for outcome 27
Measure: Mean (Standard Deviation); unit: Scale score
Arm/Group | Phase 1: 4-week Behavioral Treatment Run-in
Number analyzed (Participants) | 136
Scale score | 2.7 (1.0)

29. Other Pre Specified Outcome: Phase 1: Baseline Perceived Barriers to Healthy Eating and Physical Activity (Scale by Welsh et al., 2012)
Description: Exploratory predictor variable - phase 1 Data presented are for the total score taken as the sum of all 40 items, range 40-200. Higher total scores indicate more perceived barriers.
Time Frame: Baseline
Population: mITT analysis was planned to include all participants who provided at least one post-baseline weight measurement (N=139 out of 147). We could not include an additional 4 participants due to missing items on the scale
Measure: Mean (Standard Deviation); unit: Scale score
Arm/Group | Phase 1: 4-week Behavioral Treatment Run-in
Number analyzed (Participants) | 135
Scale score | 112.7 (25.4)

30. Other Pre Specified Outcome: Phase 1: Baseline Weight Efficacy Life-Style Questionnaire (WEL)
Description: Exploratory predictor variable - phase 1
  Weight Efficacy Life-Style Questionnaire (WEL), sum of 8 items, range 0-80, higher scores indicate greater weight-related self-efficacy
Time Frame: Baseline
Population: as for outcome 27
Measure: Mean (Standard Deviation); unit: Scale score
Arm/Group | Phase 1: 4-week Behavioral Treatment Run-in
Number analyzed (Participants) | 136
Scale score | 44.4 (16.8)

31. Other Pre Specified Outcome: Phase 1: Baseline SCI Exercise Self Efficacy Scale (ESES)
Description: Exploratory predictor variable - phase 1 SCI Exercise Self Efficacy Scale (ESES) total score, sum of 10 items, range 10-40, higher scores indicate greater exercise-related self-efficacy
Time Frame: Baseline
Population: as for outcome 27
Measure: Mean (Standard Deviation); unit: Scale score
Arm/Group | Phase 1: 4-week Behavioral Treatment Run-in
Number analyzed (Participants) | 136
Scale score | 30.6 (5.3)

32. Other Pre Specified Outcome: Phase 1: Randomization Ball and Crawford Social Support Scale
Description: Exploratory predictor variable - phase 1
  Four subscales: positive social support for eating, negative social support for eating, positive social support for exercise, and negative social support for exercise were scored separately for family and for friends. Participants rated these individuals support during the 4-week BT run-in. Participants were instructed not to answer items if not applicable. Each subscale has a range of 1-5 with higher scores indicating more positive/negative social support.
Time Frame: Randomization (week 0)
Population: mITT analysis was planned to include all participants who provided at least one post-baseline weight measurement (N=139 out of 147). Participants were instructed not to answer items if not applicable to their household/lifestyle, resulting in fewer ppts completing this scale.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Phase 1: 4-week Behavioral Treatment Run-in
Number analyzed (Participants) | 118
score on a scale
  positive eating support from family | 2.8 (1.2)
  negative eating support from family | 2.4 (0.9)
  positive exercise support from family | 2.1 (1.0)
  negative exercise support from family | 1.2 (0.4)

33. Other Pre Specified Outcome: Phase 1: Baseline Food Addiction Using the Yale Food Addiction Scale (YFAS)
Description: Exploratory predictor variable - phase 1
  The YFAS symptom count (continuous outcome) total score was used for the present data, symptom score range 0-11, higher scores indicate more food addiction symptoms
Time Frame: Baseline
Population: mITT analysis was planned to include all participants who provided at least one post-baseline weight measurement (N=139 out of 147). Additional missing data were attributable to missing item responses
Measure: Mean (Standard Deviation); unit: Symptom count
Arm/Group | Phase 1: 4-week Behavioral Treatment Run-in
Number analyzed (Participants) | 122
Symptom count | 2.4 (2.4)

34. Other Pre Specified Outcome: Phase 1: The Reinforcing Efficacy of High- and Low-calorie Food
Description: Exploratory predictor variable - phase 1 Questionnaire version of the relative reinforcing value of food computer task in which participants were asked how many servings of a preferred snack food they would consume in 1 week if they had access to no other snack foods for that week and could not stockpile for a later date. They complete this question at different price levels of the food and the reported score is the elasticity of demand which is the slope of the relationship between price (log) and number of servings that the person would purchase. Scores typically range between 0 and -2, though lower scores are theoretically possible. More negative values indicate larger reductions in purchasing of the snack food for each increase in price.
Time Frame: Baseline
Population: mITT analysis was planned to include all participants who provided at least one post-baseline weight measurement (N=139 out of 147). We could not include an additional 9 participants due to missing items on the scale
Measure: Mean (Standard Deviation); unit: (log)dollar/purchased serving
Arm/Group | Phase 1: 4-week Behavioral Treatment Run-in
Number analyzed (Participants) | 130
(log)dollar/purchased serving
  High energy density snack | -0.99 (0.21)
  Low energy density snack | -1.03 (0.21)

35. Other Pre Specified Outcome: Phase 1: Baseline Sleep Hours Survey
Description: Exploratory predictor variable - phase 1
  Average hours slept per night, including weekday and weekend nights, potential range 0 - 24, higher scores indicate more sleep
Time Frame: Baseline
Population: as for outcome 27
Measure: Mean (Standard Deviation); unit: hours slept per night
Arm/Group | Phase 1: 4-week Behavioral Treatment Run-in
Number analyzed (Participants) | 136
hours slept per night | 7.0 (1.0)

36. Other Pre Specified Outcome: Phase 1: Baseline Perceived Stress Scale
Description: Exploratory predictor variable - phase 1
  Total score on the Perceived Stress Scale, sum of 10 items, range 0-40, higher scores indicate more perceived stress
Time Frame: Baseline
Population: as for outcome 27
Measure: Mean (Standard Deviation); unit: Scale score
Arm/Group | Phase 1: 4-week Behavioral Treatment Run-in
Number analyzed (Participants) | 136
Scale score | 15.8 (6.9)

37. Other Pre Specified Outcome: Phase 1: Baseline Anxiety as Measured by the GAD-7
Description: Exploratory predictor variable - phase 1 Anxiety as measured by the GAD-7, sum of 7 items, range 0-28, higher scores indicate more anxiety
Time Frame: Baseline
Population: as for outcome 29
Measure: Mean (Standard Deviation); unit: Scale score
Arm/Group | Phase 1: 4-week Behavioral Treatment Run-in
Number analyzed (Participants) | 135
Scale score | 4.4 (4.5)

38. Other Pre Specified Outcome: Phase 1: Baseline General Mindfulness and Acceptance as Measured Using the Philadelphia Mindfulness Scale
Description: Exploratory predictor variable - phase 1
  Two separate subscales were scored: mindful awareness and acceptance, range 1-5 for both subscales. Higher scores indicate more awareness or acceptance.
Time Frame: Baseline
Population: as for outcome 27
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Phase 1: 4-week Behavioral Treatment Run-in
Number analyzed (Participants) | 136
score on a scale
  Awareness | 3.6 (3.5)
  Acceptance | 3.1 (0.8)

39. Other Pre Specified Outcome: Phase 2: Change in Blood Pressure (Systolic)
Description: Exploratory outcomes - phase 2. Systolic blood pressure
Time Frame: Week 0 (randomization) to week 24
Measure: Mean (Standard Error); unit: mm Hg
Arm/Group | Behavioral Treatment + Placebo | Behavioral Treatment + Medication
Number analyzed (Participants) | 38 | 38
mm Hg | -0.7 (1.84) | 6.6 (1.86)

40. Other Pre Specified Outcome: Phase 2: Change in Pulse
Description: Exploratory outcomes - phase 2. Pulse
Time Frame: Week 0 (randomization) to week 24
Measure: Mean (Standard Error); unit: BPM
Arm/Group | Behavioral Treatment + Placebo | Behavioral Treatment + Medication
Number analyzed (Participants) | 38 | 38
BPM | 0.09 (1.56) | 3.96 (1.50)

41. Other Pre Specified Outcome: Phase 2: Change in Triglycerides
Description: Exploratory outcomes - phase 2
Time Frame: Week 0 (randomization) to week 24
Measure: Mean (Standard Error); unit: mg/dL
Arm/Group | Behavioral Treatment + Placebo | Behavioral Treatment + Medication
Number analyzed (Participants) | 38 | 38
mg/dL | -9.00 (7.45) | -16.00 (7.25)

42. Other Pre Specified Outcome: Phase 2: Change in HDL and LDL Cholesterol
Description: Exploratory outcomes - phase 2. Reported here is HDL
Time Frame: Week 0 (randomization) to week 24
Measure: Mean (Standard Error); unit: mg/dL
Arm/Group | Behavioral Treatment + Placebo | Behavioral Treatment + Medication
Number analyzed (Participants) | 38 | 38
mg/dL | 3.27 (1.49) | 1.52 (1.37)

43. Other Pre Specified Outcome: Phase 2: Change in Fasting Blood Sugar
Description: Exploratory outcomes - phase 2. Fasting glucose.
Time Frame: Week 0 (randomization) to week 24
Measure: Mean (Standard Error); unit: mg/dL
Arm/Group | Behavioral Treatment + Placebo | Behavioral Treatment + Medication
Number analyzed (Participants) | 38 | 38
mg/dL | 1.00 (1.81) | -0.66 (1.93)

44. Other Pre Specified Outcome: Phase 2: Change in Appetite Ratings (Ratings of Appetite During the Past Week Using Visual Analogue Scales, Scored 0-100 mm)
Description: Exploratory outcomes - phase 2
  Appetite was rated weekly using the Control of Eating Questionnaire. Participants were asked to rate items based on their appetite in the past week. For the present analysis, "appetite" was calculated as the mean of the ratings for hunger, fullness after meals (reversed), and thoughts about wanting food. Higher scores (Range 0 - 100) indicate greater past-week appetite.
Time Frame: Week 0 (randomization) to week 24
Population: Randomized participants who completed the study (N = 71 of 76) and also completed the COEQ at week 24 (N = 65).
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Behavioral Treatment + Placebo | Behavioral Treatment + Medication
Number analyzed (Participants) | 30 | 35
mm
  Randomization | 48.5 (14.3) | 53.3 (13.8)
  Week 24 | 47.5 (16.8) | 42.7 (14.4)

45. Other Pre Specified Outcome: Phase 2: Change in Weight-related Quality of Life as Measured by the Impact of Weight on Quality of Life (IWQOL)
Description: Exploratory outcomes - phase 2
  Impact of Weight on Quality of Life (IWQOL) scale scores are transformed to a t-score ranging from 0-100 (e.g., 50 indicates the population mean with a standard deviation of 10). Higher t-scores are better. Positive values below for change in this measure represent improvement from randomization to week 24.
Time Frame: Week 0 (randomization) to week 24
Measure: Mean (Standard Error); unit: t score
Arm/Group | Behavioral Treatment + Placebo | Behavioral Treatment + Medication
Number analyzed (Participants) | 38 | 38
t score | 7.56 (2.18) | 9.77 (2.17)

46. Other Pre Specified Outcome: Phase 2: Change in Depressive Symptoms as Measured by the Patient Health Questionnaire (PHQ-9)
Description: Exploratory outcomes - phase 2
  Sum of 9 items, possible range 0-27. Lower scores are better (less depression). Negative values below for change in this measure represent improvement from randomization to week 24.
Time Frame: Week 0 (randomization) to week 24
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Behavioral Treatment + Placebo | Behavioral Treatment + Medication
Number analyzed (Participants) | 38 | 38
units on a scale | -0.68 (0.55) | -0.75 (0.54)

47. Other Pre Specified Outcome: Phase 2: Change in Physical Activity Using the Paffenbarger Physical Activity Questionnaire
Description: Exploratory outcomes - phase 2
  Outcome from this measure is activity minutes per week. Potential range 0 - 10,080 min/week. Higher scores indicate more minutes of activity per week. Positive values below for change in this measure represent improvement from randomization to week 24.
Time Frame: Week 0 (randomization) to week 24
Measure: Mean (Standard Error); unit: minutes per week
Arm/Group | Behavioral Treatment + Placebo | Behavioral Treatment + Medication
Number analyzed (Participants) | 38 | 38
minutes per week | 29.90 (34.02) | 91.85 (34.85)

ADVERSE EVENTS:
Time Frame: Time period: 4-week BT-run-in and 24-week randomized trial Adverse events are reported for all 147 participants during phase 1 (4-week run-in) and in phase 2 for the 76 participants who were identified as early non-responders and were randomly assigned to BT + phentermine or BT + placebo and the 55 early responders. Event frequencies for early responders cannot be compared directly to those of early non-responders because events were not queried systematically in the responder group.
Description: For randomized participants, side effects were queried during each study visit. Subjects also were instructed to contact study staff if they experience any AE between study visits. AEs were not queried systematically for non-randomized early responders but were tracked if reported to staff. The study physician or NP determined the severity of each AE and its possible relation to treatment using standard criteria, and the appropriate course of action for the study subject.
Groups:
- Phase 1: 4-week BT run-in: Adverse events occurring prior to randomization in the 147 participants who consented and enrolled in Phase 1 of the trial.
- Early Responders (Behavioral Treatment Alone): Early responders who lost >2% during the BT run-in continued to receive behavioral treatment alone for 24 more weeks and were not assigned to receive study medication. They were not considered part of the randomized trial and adverse events were not assessed systematically, so frequencies cannot be compared directly to the randomized groups.
Arm/Group | Phase 1: 4-week BT run-in | Behavioral Treatment + Placebo | Behavioral Treatment + Medication | Early Responders (Behavioral Treatment Alone)
All-Cause Mortality (participants affected / at risk) | 0/147 | 0/38 | 0/38 | 0/55
Serious Adverse Events (participants affected / at risk) | 0/147 | 0/38 | 0/38 | 0/55
Other Adverse Events (participants affected / at risk) | 23/147 | 27/38 | 23/38 | 20/55
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase 1: 4-week BT run-in (N=147) | Behavioral Treatment + Placebo (N=38) | Behavioral Treatment + Medication (N=38) | Early Responders (Behavioral Treatment Alone) (N=55)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 2 (2)
Anxiety (Psychiatric disorders) | 0 (0) | 2 (2) | 2 (2) | 2 (2)
Constipation (Gastrointestinal disorders) | 0 (0) | 3 (3) | 3 (4) | 0 (0)
COVID-19 infection (Infections and infestations) | 0 (0) | 2 (2) | 2 (2) | 4 (4)
Ear infection (Infections and infestations) | 1 (1) | 2 (2) | 1 (1) | 0 (0)
Headache (General disorders) | 2 (3) | 2 (2) | 6 (6) | 3 (3)
Musculoskeletal Injury (Musculoskeletal and connective tissue disorders) | 7 (9) | 4 (4) | 4 (4) | 4 (6)
Sinus infection (Infections and infestations) | 2 (2) | 4 (4) | 2 (2) | 0 (0)
Upper respiratory infection (Infections and infestations) | 7 (7) | 13 (15) | 4 (4) | 5 (5)
Reaction to COVID-19 vaccine (General disorders) | 3 (3) | 2 (2) | 1 (2) | 2 (2)
Vomiting (Gastrointestinal disorders) | 1 (1) | 2 (2) | 0 (0) | 1 (1)
Difficulty sleeping (Psychiatric disorders) | 0 (0) | 0 (0) | 3 (3) | 2 (2)
Dry mouth (General disorders) | 0 (0) | 0 (0) | 4 (6) | 0 (0)
Nausea (Gastrointestinal disorders) | 2 (2) | 0 (0) | 2 (2) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-05-05): https://cdn.clinicaltrials.gov/large-docs/48/NCT03779048/Prot_SAP_000.pdf